CLINICAL TRIAL: NCT05935059
Title: Evaluation of the Efficacy of Perioperative Administration of Tianeptine Versus Pregabalin on Acute and Chronic Post Mastectomy Pain After Breast Cancer Surgery. A Double-Blinded Randomized Controlled Trial.
Brief Title: The Efficacy of Tianeptine Versus Pregabalin on Acute and Chronic Post Mastectomy Pain After Breast Cancer Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ayman Sharawy Abdel Rahman Aboul Nasr, Principal investigator, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AP2305.501.039
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Post-mastectomy Pain Syndrome
Keywords: Breast cancer; Post mastectomy pain; chronic pain
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain | interventions — Pregabalin; Anticonvulsants; tianeptine; Antidepressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pregabalin group (group P) (Active Comparator): pregabalin group (group P) patients will receive pregabalin (Lyrica, Pfizer, NY) 50 mg with a sip of water one hour before induction of anesthesia and repeated every 8 hours for five days after surgery. The pregabalin capsules will be given to patients by nurses blinded to the study. Neither the researcher allocating the participants, nor the assessing person knew the decoding of the groups in its relation to the allocation sequence. Data will be collected by a junior pain resident blinded to the study protocol.
  Interventions: Drug: Pregabalin
- Tianeptine group (group T) (Active Comparator): Tianeptine group (group T) patients will receive Tianeptine 12.5 mg (Stablon, Servier, France)with a sip of water one hour before induction of anesthesia and repeated every 8 hours for five days after surgery. The Tianeptine capsules will be given to patients by nurses blinded to the study. Neither the researcher allocating the participants, nor the assessing person knew the decoding of the groups in its relation to the allocation sequence. Data will be collected by a junior pain resident blinded to the study protocol.
  Interventions: Drug: Tianeptine

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 50Mg Oral Capsule. Pre-operative administration of Pregabalin for prevention of Post mastectomy Pain Syndrome (PMPS)
  Other Names: Anticonvulsant
  Arms: pregabalin group (group P)
Drug: Tianeptine — Tianeptine 12.5Mg Capsules. Prevention of Post Mastectomy Pain Syndrome
  Other Names: Antidepressant
  Arms: Tianeptine group (group T)

SUMMARY:
Breast cancer is the most common malignancy among females. Nearly 40% of breast surgery patients experience moderate to severe acute postoperative pain, with severe pain persisting for more than 6 months in almost 20-50% of patients (post mastectomy pain syndrome) which is defined according to International Association for the Study of Pain (IASP) as pain which persists more than 3 months after mastectomy/lumpectomy affecting the anterior thorax, axilla, and/or medial upper arm. Different pharmacological tools have been in use for either prevention or treatment of such refractory pain syndrome with variable efficacy. The aim of this study is to assess the efficacy of the perioperative use of Pregabalin versus Tianeptine on the emergence of PMPS in female patients undergoing MRM for breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most common diagnosed malignancy among females and the 5th cause of cancer-related deaths with an estimated number of 2.3 million new cases and 685,000 deaths worldwide in 2020.

Different modalities are used for management of breast cancer including surgery, radiation therapy (RT), chemotherapy (CT), endocrine (hormone) therapy (ET), and targeted therapy. Modified Radical Mastectomy (MRM) is one of the main modalities of breast cancer treatment. It accounts for 31% of all breast surgeries. It has been reported that 40% of the females complain from moderate-to-severe pain in the immediate post-operative period after breast cancer surgery.

Acute post-mastectomy pain can cause adverse impacts on the patients as delayed discharge from post-operative recovery area, impairs pulmonary and immune functions, increases risk of ileus, thromboembolism, myocardial infarction and may lead to increased length of hospital stay. It is also an important factor leading to the development of chronic post mastectomy pain syndrome (PMPS) in almost half of the patients.

The International Association for the Study of Pain (IASP) defines PMPS as pain which persists more than 3 months after mastectomy that affects the anterior thorax, axilla, and/or medial upper arm. It is usually described as the feeling of burning, stabbing, and pulling around the treatment side. The underlying pathophysiology of PMPS is highly complicated and involves both peripheral and central sensitization. It results from injury to the peripheral nerves in the axilla or the chest wall during the dissection of axillary lymph nodes. Multiple risk factors are involved in the development of PMPS including acute postoperative pain, age < 40 years, increased BMI , diagnosis at later-stage disease, psychosocial factors (i.e., anxiety, depression, sleep disturbances, catastrophizing), preoperative pain and adjuvant therapy (chemotherapy, radiation therapy).(8)Because PMP involves issues associated not only with pain management, but also with psychosocial disruption, the assessment of each of these domains should be addressed routinely so as to enable early detection and treatment.

Different pharmacological tools have been in use for either prevention or treatment of such refractory pain syndrome with variable efficacy.

Tianeptine is a unique antidepressant and anxiolytic medication that stimulates the uptake of serotonin (5-hydroxytryptamine; 5-HT), and 5-hydroxyindoleacetic acid (5-HIAA) in brain tissue . It acts as a full agonist at the mu-type opioid receptor (MOR) , the serotonin receptor ,dopamine (D2/3) receptors and glutamate receptors .It also reduces the hypothalamic-pituitary-adrenal response to stress, and thus prevents stress-related behavioral issues.

Pregabalin is a new synthetic molecule and a structural derivative of the inhibitory neurotransmitter γ-aminobutyric acid. It is an α2-δ (α2-δ) ligand that has analgesic, anticonvulsant, anxiolytic, and sleep-modulating activities. Pregabalin binds potently to the α2-δ subunit of calcium channels, resulting in a reduction in the release of several neurotransmitters, including glutamate, noradrenaline, serotonin, dopamine, and substance P , Pregabalin has also been found to be effective at reducing acute postoperative pain The efficacy of pregabalin in treating acute postsurgical pain has been demonstrated in numerous studies. A recent meta-analysis has suggested that pregabalin, at all doses and administration regimens, has opioid-sparing effects and reduces pain scores in the postsurgical setting, at the expense of increased sedation and visual disturbances; however, the efficacy of pregabalin in providing such in various surgical categories remains uncertain, and it is not known whether the risk: benefit ratio is greater for certain surgical categories The aim of this study is to assess the efficacy of the perioperative use of Pregabalin versus Tianeptine on the emergence of PMPS in female patients undergoing MRM for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer female patients.
2. ASA class II and III.
3. Age ≥ 18 and ≤ 60 Years.
4. Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.
5. Type of surgery; elective breast cancer surgery (either modified radical mastectomy or conservative breast surgery) combined with axillary dissection.

Exclusion Criteria:

1. Patient refusal.
2. Age <18 years or >65 years.
3. BMI <20 kg/m2 and >35 kg/m2.
4. Known sensitivity or contraindication to drugs used in the study (Pregabalin , Tianeptine , NSAIDs, or morphine ).
5. History of psychiatric disorders or history of major depression.
6. History of chronic pain that necessitates morphine at a daily dose of 30 mg or more (or equivalent opioids).
7. history of gapabentenoids or antidepressant intake in the preceding three months.
8. Major medical conditions.
9. Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
the percentage of patients who developed Post Mastectomy Pain Syndrome (PMPS) | 6 months
  The Percentage of patients developing Post Mastectomy Pain Syndrome (PMPS)

SECONDARY OUTCOMES:
Changes and stability in Mean Arterial Blood Pressure (MAP) | every 15 minutes during the surgery then at 1, 2, 4, 8, 12, 16, 20 and 24 hours postoperatively
  Change in Mean Arterial Blood Pressure (MAP) in mmHg
Changes and stability in Heart Rate (HR) | every 15 minutes during the surgery then at 1, 2, 4, 8, 12, 16, 20 and 24 hours postoperatively
  Change in heart rate (HR) in beat\min
Total amount of fentanyl consumed intraoperative | Time of surgery
  the rescue analgesia will be administered intra-operative by fentanyl IV and the total fentanyl used will be recorded and compared between the groups
1st time opioids requested post-operative. | 24 hours after the surgery
  In case of postoperative pain recorded, rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the patient VAS Score ≥ 4. The total amount of morphine given in 24 hours will be recorded for both groups
Total amount of morphine consumed postoperatively | 24 hours after the surgery
  The total 24-hour morphine consumption will be recorded for every patient post operative.
The degree of postoperative sedation according to Ramsay scores. | 24 hours
  Sedation will be assessed with Ramsay score (1 = anxious or restless or both; 2 = cooperative, orientated, and tranquil; 3= responding to commands; 4 = brisk response to stimulus; 5 = sluggish response to stimulus; and 6 = no response to stimulus). A Ramsay score of 5 or 6 will be considered excessively high sedation levels; a Ramsay score of 2 to 4 will be considered adequate sedation levels needing observation; a Ramsay score of 1 will be considered inadequate or insufficient sedation Levels
Postoperative nausea and vomiting (PONV). | 24 hours
  Postoperative nausea and vomiting (PONV) will be rated on a four-point verbal scale; (none =no nausea, mild =nausea but no vomiting, moderate=vomiting one attack, severe =vomiting >one attack). 0.1 mg/kg of IV ondansetron will be given to patients with moderate or severe postoperative nausea and vomiting.
Severity of PMPS according to Grading system for neuropathic pain (GSNP) | 6 motnths
  Neuropathic pain will be evaluated according to the Grading System for Neuropathic Pain (GSNP). Positive neuropathic cases are those with GSNP 3 (probable) or GSNP 4 (definite) i.e. GSNP ≥ 3 . Grading system for neuropathic pain (GSNP) is as follows: Grade 1 (unlikely), Grade 2 (possible), Grade 3 (probable), and Grade 4 (definite )

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Sharawy Abdel Rahman Aboul Nasr, MD, Principal Investigator — National Cancer Institute Cairo University
Locations (1):
- National Cancer Institute Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Dhankhar R, Vyas SP, Jain AK, Arora S, Rath G, Goyal AK. Advances in novel drug delivery strategies for breast cancer therapy. Artif Cells Blood Substit Immobil Biotechnol. 2010 Oct;38(5):230-49. doi: 10.3109/10731199.2010.494578. PMID 20677900
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Capuco A, Urits I, Orhurhu V, Chun R, Shukla B, Burke M, Kaye RJ, Garcia AJ, Kaye AD, Viswanath O. A Comprehensive Review of the Diagnosis, Treatment, and Management of Postmastectomy Pain Syndrome. Curr Pain Headache Rep. 2020 Jun 11;24(8):41. doi: 10.1007/s11916-020-00876-6. PMID 32529416
- [Background] Samuels BA, Nautiyal KM, Kruegel AC, Levinstein MR, Magalong VM, Gassaway MM, Grinnell SG, Han J, Ansonoff MA, Pintar JE, Javitch JA, Sames D, Hen R. The Behavioral Effects of the Antidepressant Tianeptine Require the Mu-Opioid Receptor. Neuropsychopharmacology. 2017 Sep;42(10):2052-2063. doi: 10.1038/npp.2017.60. Epub 2017 Mar 17. PMID 28303899
- [Background] Reyad RM, Omran AF, Abbas DN, Kamel MA, Shaker EH, Tharwat J, Reyad EM, Hashem T. The Possible Preventive Role of Pregabalin in Postmastectomy Pain Syndrome: A Double-Blinded Randomized Controlled Trial. J Pain Symptom Manage. 2019 Jan;57(1):1-9. doi: 10.1016/j.jpainsymman.2018.10.496. Epub 2018 Oct 22. PMID 30359684